CLINICAL TRIAL: NCT04092049
Title: Effect of Chewing Lollipop on Gastric Emptying
Brief Title: Lollipop on Gastric Emptying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: XJH-A-20190916
Record Dates: First submitted 2019-09-15; First posted 2019-09-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Gastric Emptying

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lollipop (Experimental)
  Interventions: Other: lollipop
- control (No Intervention)

INTERVENTIONS:
Other: lollipop — chewing lollipop for 10 minutes
  Arms: lollipop

SUMMARY:
To investigate the effect of chewing lollipop on gastric volume and gastric emptying in healthy volunteers drinking water.

ELIGIBILITY:
Inclusion Criteria:

* volunteer aged 18 years-45 years old
* volunteer with a body mass index between 18 and 28 kg/m2

Exclusion Criteria:

* those with history of diabetes mellitus
* those with gastric diseases
* those with history of gastro-intestinal surgery
* those with history of smoking
* those with use of gastric mobility medicines
* those with pregnancy or breeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2019-12-22 (Actual)

PRIMARY OUTCOMES:
half time of gastric emptying | from drinking water to gastric volume return to half of top volume before drinking water,on an average of 2 hours

SECONDARY OUTCOMES:
time of gastric emptying | from drinking water to gastric volume return to baseline before drinking water,on an average of 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual Data of primary outcome and secondary outcome will be shared

REFERENCES:
- [Result] Bouvet L, Loubradou E, Desgranges FP, Chassard D. Effect of gum chewing on gastric volume and emptying: a prospective randomized crossover study. Br J Anaesth. 2017 Nov 1;119(5):928-933. doi: 10.1093/bja/aex270. PMID 29077816